CLINICAL TRIAL: NCT02743507
Title: The Impact of the Bundled Payments for Care Improvement Program on Quality and Costs of Care
Brief Title: The Impact of Bundled Payments on Quality and Cost of Care
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Amol Navathe, Amol Navathe, MD, PhD, University of Pennsylvania
Other Study IDs: 824812
Record Dates: First submitted 2016-04-08; First posted 2016-04-19 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis; Chronic Obstructive Pulmonary Disease; Pneumonia
MeSH Terms: conditions — Osteoarthritis; Pulmonary Disease, Chronic Obstructive; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bundled payment is a new payment reform that encourages health care providers to improve quality and contain costs of care. These arrangements are being rapidly expanded across the country, but evidence about their impact are lacking. This study will use Medicare claims data to evaluate the effect of participation in a large Medicare bundled payment program on the quality and costs of care for common medical and surgical conditions.

DETAILED DESCRIPTION:
The overall objective is to examine the effects of the Bundled Payments for Care Improvement (BPCI) Model 2 on the quality and costs of care for conditions related to seven of the ten Medicare severity disease-related groups (MS-DRGs) most commonly selected by program participation. Five of these are surgical (major joint replacement of the lower extremity; double joint replacement of the lower extremity; revision of the hip or knee, hip and femur procedures except major joint; lower extremity and humerus procedure except hip, foot, and femur) and two are medical (simple pneumonia and respiratory infections; chronic obstructive pulmonary disease, bronchitis/asthma). These MS-DRGs represent two larger service lines: orthopedics and pulmonary. For each of these seven MS-DRGs, the team will first describe characteristics of provider organizations participating in bundled payment arrangements, including geographic characteristics and clinical volume. We will subsequently empirically test the effect of bundled payment arrangements on quality outcomes and costs of care for these conditions. Additionally, the team will examine any spillover effects that occur within the service lines that contain these seven MS-DRGs.

ELIGIBILITY:
Inclusion Criteria:

* Provider organizations that participate in model 2 of the BPCI program, accept bundled payment for the ten most common MS-DRGs, and have at least ten or greater episodes in each of the MS-DRGs.

Exclusion Criteria:

* Provider organizations who participated in the BPCI program, but do not meet inclusion criteria will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population consists of a subset of provider organizations who participated in CMS's BPCI bundled payment program. From this group, the team will focus on provider organizations that participated in the largest model within the BPCI program (model 2) and accepted bundled payment for the ten most common MS-DRGs.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12-31 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Unplanned readmission rates | Up to 90 days
  The study team will analyze changes in unplanned admission rates at 30, 60, and 90 days post-discharge.
Emergency department utilization rates for patients post-discharge | 12 months
  The study team will analyze post-discharge emergency department utilization without re-hospitalization in patients with the specific 10 MS-DRGs to test the effect of bundled payment arrangements on quality outcomes and costs of care for these conditions.
All-cause mortality | 12 months
  The study team will analyze all cause mortality in patients with the specified 10 MS-DRGs.

SECONDARY OUTCOMES:
Total Medicare per patient per episode | 12 months
  The study team will analyze total Medicare episode spending for individual patients to test the effect of bundled payment arrangements on quality outcomes and costs of care for these conditions.
Medicare spending per patient for the initial hospitalization | 12 months
  The study team will analyze Medicare spending for initial hospitalization and for services during the initial post-hospitalization period to test the effect of bundled payment arrangements on quality outcomes and costs of care for these conditions.

IPD SHARING:
Plan to Share IPD: No